CLINICAL TRIAL: NCT01680029
Title: A Clinical Investigation to Evaluate the Safety and Performance of the PBASE-system When Used in the Treatment of Acute Migraine Episodes of Moderate to Severe Intensity
Brief Title: PBASE-system Acute Migraine Clinical Investigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too slow recruitment rate
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM001
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Acute Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PBASE-system 2.0 (Experimental)
  Interventions: Device: PBASE-system 2.0

INTERVENTIONS:
Device: PBASE-system 2.0

SUMMARY:
To evaluate the performance and safety of the PBASE-system when used in the treatment of acute migraine episodes of moderate to severe intensity. The study will evaluate the effect of treatment on migraine pain and symptoms during an acute attack and also any long-term effect.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to participation in the clinical investigation
* Male or female aged between 18 and 65 years
* Diagnosed as suffering from migraine with or without aura according to IHS classification (ICHD-II)
* Reported history of 2 to 6 migraine episodes per month during previous 3 months, confirmed during a prospective baseline period of one month
* Reported history of no less than 50% of migraine episodes involving moderate or severe pain intensity, confirmed during a prospective baseline period of one month
* Reported history of at least 48 hours of freedom from headache between migraine attacks, confirmed during a prospective baseline period of one month
* Reported history of the majority of untreated migraine attack durations lasting 8 hours or more
* Onset of migraine headache occured before age 50
* Reported history of migraine for more than one year
* Able and willing to maintain current preventive headache medication regimen(s) (no change in type, frequency or dose) from baseline screening visit to 2 weeks post-treatment
* Able to understand and complete the electronic diary
* Experiencing an acute migraine attack of moderate to severe pain intensity at the time of treatment
* Treatment is possible within 5 hours of migraine onset

Exclusion Criteria:

* Reported history of 15 or more headache days per month (i.e. headaches of any kind), confirmed during a prospective baseline period of one month
* Reported frequency of non-migraine headaches exceeding 6 days per month, confirmed during a prospective baseline period of one month
* Unable to distinguish between migraine headaches and other headache types at the onset of a migraine attack
* Treatment with Botox received within 6 months of the screening visit, or between the screening and treatment visit
* Previously treated with an implantable stimulator or any implantable devices in the head and/or neck
* Diagnosed as having a pronounced anterior septal deviation
* History of sinus surgery, transphenoidal surgery for pituitary or other lesions or CSF rhinorrhea
* Fitted with a pacemaker /defibrillator
* Previously treated with radiation to the face
* Ongoing bacterial infection in the nasal cavity
* History of nose bleeds (epistaxis)
* Ongoing malignancy in the nasal cavity
* Concomitant condition that could cause excessive bleeding
* Known allergy to polyvinylchloride,the material used for fabrication of the balloon part of Catheter A100, or medicinal liquid paraffin
* Concurrent condition or risk of non-compliance that, in the investigator's opinion, may affect the interpretation of performance or safety data or which otherwise contraindicates participation in a clinical investigation
* Any change in migraine prophylaxis between the screening and treatment visit
* Women of childbearing potential who is pregnant or at risk of becoming pregnant prior to or during the treatment phase
* Participation in a clinical research study within 3 months of enrolment or planned participation at any time during this clinical investigation
* Considered to meet the definition of vulnerable in the Investigator's opinion
* Headache or migraine episode within the 48 hours prior to treatment
* PRN (as required) or acute migraine medication(s) taken within the 48 hours prior to treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01

PRIMARY OUTCOMES:
Headache relief | 2 hours post-initiation of treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Glasgow
  - London
  - Stoke-on-Trent